CLINICAL TRIAL: NCT00159952
Title: Effect of Hyperglycemia in PAI-1 Activity and the Relationship With Outcome in Severe Sepsis and Septic Shock
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Policlinico Hospital (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Luciano Gattinoni, Policlinico Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3133; Lilly F1K0020; MIUR 2004060419
Record Dates: First submitted 2005-09-07; First posted 2005-09-12 (Estimated); Last update posted 2013-11-27 (Estimated); Status verified 2009-02

CONDITIONS: Severe Sepsis; Septic Shock
Keywords: Sepsis; Septic shock; Hyperglycemia; Fibrinolysis; PAI 1
MeSH Terms: conditions — Sepsis; Shock, Septic; Hyperglycemia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Active Comparator)
  Interventions: Procedure: intensive insulin therapy

INTERVENTIONS:
Procedure: intensive insulin therapy — control: glycemia will be controlled with insulin administration when higher than 215 mg/dL.
  treatment: glycemia will be controlled with be controlled with insulin administration when higher than 110 mg/dL

SUMMARY:
The purpose of this study is to determine the effect of the intensive insulin therapy on coagulation and fibrinolysis in patients affected by severe sepsis and septic shock. As a secondary endpoints the investigators will determine the effect of intensive insulin therapy on organ dysfunction and mortality of these patients.

DETAILED DESCRIPTION:
BACKGROUND

The treatment of the sepsis can be done at three different level:

1. Etiologic therapy. The eradication of the infectious agent is the primary end-point. An appropriate surgical treatment and antibiotic therapy are the key of the etiologic therapy.
2. Symptomatic therapy. It is the traditional approach in the Intensive Care Unit. It involves to correct the symptomatic issues that can lead to the death of the patients, buying the time necessary for the action of the etiologic and the pathogenic therapy. The key point of the symptomatic therapy are: a) an adequate expansion of the volemia and the use of cardiovascular-acting drugs, for the maintenance of an adequate cardiocirculatory homeostasis. Recently it has been demonstrated that an early aggressive haemodynamic therapy direct to maintain a mixed venous Oxygen Saturation above 70% improved the mortality compared with a standard approach (3); b) apply a mechanical ventilation adequate for the maintenance of the respiratory homeostasis. In fact it has been recently shown an increased survival rate in patients treated with low tidal volume ventilation strategy compared to standard strategy.
3. Pathogenic therapy. It consists to block the inflammatory and/or coagulation pathway at different level. In the last 30 years a number of report studied different approach (anti-endotoxin antibodies, anti-TNF antibodies, anti-IL6 antibodies, treatment with high doses of corticosteroid, etc.). While all these approaches showed an efficacy in experimental settings when given preventively, most of them have no effect in phase 3 clinical trial. This discrepancy may be explained considering: 1) the system can be considered chaotic, with riddance and interdependency of the response; 2) in the clinical studies the treatment was applied after the development of the sepsis, when the inflammatory and coagulation systems are still largely activated.

Three study has recently demonstrated a benefit in survival:

1. The treatment with low-dosage corticosteroids in patients non-responders to ACH stimulation test (5). This is a substitutive therapy. It is important to note that the treatment with high dosage corticosteroids to block completely the inflammatory response is not effective (6).
2. The treatment with recombinant activated Protein C (7) did increased the relative survival rate by 20%. Of note the activated Protein C is the only molecule with three main mechanisms of action: anticoagulatory, antiinflammatory and profibrinolytic.
3. In a recent study in post-surgical patients it has been shown a significant improvement in survival in patients treated with a a tight glycemic control within 80 and 110 mg/dL compared to those in which the glycemia was corrected only when reaching higher level (>215 mg/dL) (8).We still lack a definitive explanation for these findings, and the discussion is mainly on the relative roles of glycemia per se versus insulin therapy per se.

However, looking at the overall scenario, some issues are of note:

1. We know that a complete block of the inflammatory reaction or a complete block of the coagulation cascade do not improve outcome in septic patients
2. The activated Protein C is the molecule with the highest spectrum of action, in particular is the only molecule within the numerous molecules tested with pro-fibrinolytic activity
3. We know that higher glycemia per se does greatly increase the PAI production (the molecule which inhibits the fibrinolysis).
4. The septic patients primarily die because of multiple organ dysfunction which is in part due to a widespread microthrombosis.

A possible unifying hypothesis is that the improved outcome observed with activate Protein C and with the tight glycemic control is due to the maintenance of a physiologic fibrinolysis. This hypothesis has never been tested and if proved could open interesting therapeutical approaches in the septic patients exposed to the high mortality risk.

OBJECTIVES: The primary end-point is the evaluation of the activation/deactivation of the fibrinolytic system in the two-randomization groups.

STUDY DESIGN: This study is a multicenter, randomized, Phase 2/3 study of adult patients with severe sepsis and septic shock. We will enroll a total of approximately 80 adult patients.

TREATMENTS ADMINISTERED

1. Control: glycemia will be controlled with insulin administration when higher than 215 mg/dL.
2. Treatment: glycemia will be controlled with be controlled with insulin administration when higher than 110 mg/dL.

RANDOMIZATION: The patients enrolled will undergo a block-randomization by center in two arms and stratified according to the clinical decision of the caring physician to use or not use the activated Protein C.

DATA COLLECTION: The clinical variables and the biochemical variables of fibrinolysis, coagulation, contact phase and pro-inflammatory cytokines will be recorded daily for the first 7 days, each second day until the 14 days and the each fifth until the end of the study (28th day, or dimission/death if before).

At Baseline:Demographic data

Every 24 hours:

1. Simplified Acute Physiology Score II (SAPS II) (9). The Simplified Acute Physiology Score assesses the severity of illness on the basis of 12 physiological variables; age, the type of admission (urgent or nonurgent) and 3 variables related to the underlying disease. Scores can range from 0 to 194; higher scores are correlated with a higher risk of death during hospitalization
2. SOFA (Sepsis-related Organ Failure Assessment) (10). It is an index of multi-organ dysfunction (range 0-24).
3. Ramsey scale (11). It is an index of level of sedation (range 1-6).
4. Respiratory, circulatory and biochemical of variables for monitoring the organs dysfunction (4).

The main biochemical variables collected are:

* Fibrinolytic system:

  1. PAI-1 activity
  2. PAI- 1 antigen
  3. tPA antigen
  4. Plasmin-antiplasmin complex (PAP)
  5. D-Dimer fragment
  6. Polymorphism 4G/5 of the PAI-1 gene
* Final phase pf the coagulation pathway

  1. Thrombin-antithrombin complex (TAT)
  2. Prothrombin fragment F1 + 2
* Contact system

  1. Activated Factor XII (FXIIa)
  2. Metabolism of endogenous bradykinin
  3. Polymorphism insertion/deletion of the gene of angiotensin converting enzyme
* Inflammation

  1. C reactive protein (CRP)
  2. Interleukin-6 (IL-6)
  3. Tumor necrosis factor (TNF)
  4. C3a
  5. SC5b-9

SAFETY ASPECTS AND SEVERE ADVERSE EVENTS (SAE) REPORTING: GCP rules will be strictly applied, including timely reporting to the study coordination within 48 hours from their occurrence of the SAEs not included in the efficacy end-points. Clinical investigators and nurses of each of the participating centers will be instructed to monitor specifically and to document the adverse events more likely to be associated with the study treatment.

STATISTICAL ASPECTS: we plan to enroll 80 septic patients in the ICU related with the participating research units. This size will allow showing an average difference of 30% of fibrinolysis biochemical parameters (alfa = 0.05, 1-beta = 0.80).

ADMINISTRATIVE, LEGAL, ETHICAL ISSUES: This study is designed by our collaborative group, which has been active over the last ten years in conducting clinical trials in intensive care. The study has been planned and is managed independently, and the clinicians who take active part in the study do not receive economic incentives. The Ely Lilly Italia Spa will provide a financial support for performing the laboratory tests required in studying the fibrinolysis. It is important to emphasize that we are comparing the effects of two different strategies of glycemic control on the fibrinolysis. The Ely Lilly interest in the study is only scientific, as, if we could show the importance of the fibrinolysis in sepsis, this could elucidate one of the putative mechanisms of activated Protein C action. This study is also partially funded by a grant of the Ministry of University and research (COFIN 2004).

The data which are produced belong to the study group, who ensures their publication and their availability for public authorities.

All data related to the patients included in the study are treated in strict compliance with the Italian Laws related to privacy 675/1996.

The informed consent for the patients will be administered as soon as and every time the clinical conditions of the same patients are compatible with the procedure, thus following the provisions set forth by the ICH-GCP guidelines (13), and confirmed by the most recent European Directive 2001/20/CE Decreto Legislativo 211 24/06/2003. It is worth recalling that there is no legal basis for requiring the consent to a relative of the patient.

REFERENCES

1. Gattinoni L, Vagginelli F, Taccone P, Carlesso E, Bertoja E, Sepsis: state of the art. Minerva Anestesiologica 2003; 69: 17-28.
2. Salvo I, de Cian W, Musico M. Langer M, Piadina R, Wolfer A, et al. The Italian SEPSIS study: preliminary results on the incidence and evolution of SIRS, sepsis, severe sepsis and septic shock. Intensive Care Medicine 1995; 21 Suppl. 2:S244-249.
3. Rivers E, Nguyen B, Havstad S, Ressler J, Muzzin A, Knoblich B, et al. Early goal-directed therapy in the treatment of severe sepsis and septic shock. The New England Journal of Medicine 2001; 345: 1368-1377
4. Ventilation with lower tidal volumes as compared with traditional tidal volumes for acute lung injury and the acute respiratory distress syndrome. The New England Journal of Medicine 2000; 342: 1301-1308
5. Annane D, Sibille V, Charpentier C, Bollaert PE, Francois B, Korach JM , et al. Effect of treatment with low doses of hydrocortisone and fludrocortisone on mortality in patients with septic shock. JAMA 2002; 288: 862-871
6. Bone RC, Fischer CJJ, Clemer TP, Slotman GJ, Metz CA Balk RA. A controlled clinical trial of high-dose methyl-prednisolone in the treatment of severe sepsis and septic shock. The New England Journal of Medicine 1987; 317: 653-658
7. Bernard GR, Vincent JL, Laterre PF, La Rosa SP, Dhainaut JF, Lopez-Rodriguez A, et al. Efficacy and safety of recombinant human activated protein C for severe sepsis. The New England Journal of Medicine 2001; 344:699-709
8. Van de Berghe G, Wouters P, Weekers F, Verwaest C, Brunynckx F, Schets M, et al. Intensive insulin therapy in the critically ill patients. New Engl j med 2001; 345:1359-1367
9. Knaus WA, Draper EA, Wagner DP, Zimmerman JE, APACHE II: a severity of disease classification system. Crit Care Med 1985; 13: 818-829
10. Vincent JL, de Mendonca A, Contraine F, Moreno R, Takala J, Suter PM, Sprung CL, Colardyn F, Blecher S, Use of the SOFA score to assess the incidence of organ dysfunction/failure in intensive care units: results of a multicenter prospective study. Working group on "sepsis-related problems" of the European Society of Intensive Care Medicine. Crit Care Med 1998; 26:1793-800
11. Ramsay MAE, Savege TM, Simpson BRJ et al.: Controlled sedation with alphaxalone-alphadolone. Br Med J 1974; 2: 656-659
12. Dhainaut JF, Yan SB, Cariou A, Mira JP. Soluble thrombomodulin, plasma-derived unactivated protein C, and recombinant human activated protein C in sepsis. Crit Care Med 2002 May; 30 (5 Suppl): S318-24
13. Guidelines for Good Clinical Practice, par. 4.8. ICH Steering Committee meeting. 1 May 1996.

ELIGIBILITY:
Inclusion Criteria:

Patients with sepsis, severe sepsis and sepsis shock defined as follows:

Sepsis:

Systemic response to infection with two or more of the following conditions:

* Body temperature<36° or >38°
* Heart rate >90 bpm
* Respiratory rate >20 bpm or PaCO2<32 torr
* White cells count>12000 mm3 or <4000 mm3 or a differential count showing>10% of immature neutrophiles

Severe sepsis:

* Sepsis associated to a organ dysfunction.

Sepsis shock:

* Sepsis associated to hypotension despite adequate fluid resuscitation, with hypoperfusion including lactic acidosis, oliguria and acute alteration of consciousness. The hypotension does not need to be present in patients treated with inotropic or vasoactive drugs.

Exclusion Criteria:

* Age below 16 years
* Patients with hematologic malignancy or bone marrow transplant
* Patients with type I diabetes
* Patients with expected early death because of underlying disease.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2004-11; Primary Completion 2007-03 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
The primary end-point is the evaluation of the activation/deactivation of the fibrinolytic system in the two randomization group | At Baseline and every 24 hour

SECONDARY OUTCOMES:
To evaluate the different organ dysfunctions (pulmonary, hepatic and volemic status) | 28 days survival
The effect of the treatment | 28 days survival

CONTACTS AND LOCATIONS:
Overall Officials: Luciano Gattinoni, MD, Principal Investigator — Policlinico Hospital of Milan
Locations (3):
- Italy (3):
  - Hospital "S.Paolo", Milan
  - Policlinico Hospital, Milan
  - Hospital "S.Gerardo", Monza

REFERENCES:
- [Derived] Savioli M, Cugno M, Polli F, Taccone P, Bellani G, Spanu P, Pesenti A, Iapichino G, Gattinoni L. Tight glycemic control may favor fibrinolysis in patients with sepsis. Crit Care Med. 2009 Feb;37(2):424-31. doi: 10.1097/CCM.0b013e31819542da. PMID 19114908